CLINICAL TRIAL: NCT01352039
Title: A Phase III, Non-inferiority, Randomized, Double-blind Trial Comparing Eurofarma Unfractionated Sodium Heparin 5,000 IU to APP Pharmaceuticals Unfractionated Sodium Heparin 5,000 IU in the Thromboprophylaxis of Geriatric Patients Who Underwent Hip Fracture Surgery.
Brief Title: A Non-inferiority Study Comparing Two Heparin Sodium Preparations in Hip Fracture Surgery
Acronym: HEP-SC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EF098 - HEP-SC
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Hip Fracture Surgery
Keywords: Heparin Sodium; Thromboprophylaxis; Hip Fracture Surgery.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparin Sodium - Eurofarma (Experimental)
  Interventions: Biological: Heparin Sodium - Eurofarma
- Heparin Sodium - APP Pharmaceuticals (Active Comparator)
  Interventions: Biological: Heparin Sodium - APP Pharmaceuticals

INTERVENTIONS:
Biological: Heparin Sodium - Eurofarma — Heparin Sodium will be given during 5 to 7 days each 8 hours on dosis 5,000 UI
  Arms: Heparin Sodium - Eurofarma
Biological: Heparin Sodium - APP Pharmaceuticals — Heparin Sodium will be given during 5 to 7 days each 8 hours on dosis 5,000 UI
  Arms: Heparin Sodium - APP Pharmaceuticals

SUMMARY:
The primary objective and endpoints of the study is compare the efficacy of two products containing heparin sodium, evaluating if the formulation produced by Eurofarma can be considered non-inferior to the reference product.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the efficacy of unfractionated heparin sodium of porcine origin (Eurofarma) in the prophylaxis of VTE relative to unfractionated heparin sodium of porcine origin from APP Pharmaceuticals. The primary endpoint will be the frequency of DVT determined by Doppler ultrasound (DUS).

ELIGIBILITY:
Inclusion Criteria:

In order to be enrolled in this study, eligible patients must meet all criteria below:

* ICF signing;
* Aged 60 to 85 years old;
* Indication of hip orthopedic surgery due to fracture occurred within the last 5 days;
* Normal coagulation profile or with alterations up to 25% of normal values.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible for the study:

* Previous hip surgery;
* Fracture secondary to the presence of metastasis;
* Recent traumatic brain, thoracic, or abdominal injury (up to 30 days before study start);
* Recent occurrence (up to 30 days before study start) of cerebrovascular accident;
* Serum concentration of hemoglobin below 9 g/dL;
* Prior occurrence (in the last 5 years) of confirmed or suspected thromboembolic event;
* Occurrence of major bleeding in the last 6 months (any spontaneous gastrointestinal bleeding; central nervous system bleeding; massive epistaxis, or gum bleeding; gross hematuria, or vaginal bleeding);
* Confirmed or suspected blood dyscrasia;
* Diagnosis of neoplasm other than in situ in the last 24 months or any active neoplasm (neoplasms in situ do not prevent patient from participating);
* Liver or kidney failure;
* Clinically significant gastrointestinal cardiovascular, neurological disease, or laboratory abnormalities, which at the investigator's opinion, may interfere with individual's participation in the study or with assessment of individual's response to treatment;
* Hypersensitivity to heparin;
* Previous use (15 days before study start) of oral anticoagulants or expected use during the study (see Appendix B);
* Recent participation (previous 12 months) in a clinical trial.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The Primary endpoint will be frequency of deep venous thrombosis (DVT) determined by Doppler ultrasound (DUS). | 6 months

SECONDARY OUTCOMES:
The Secundary endpoint will be proximal and distal DVT | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Centro de Pesquisa Clínica da Santa Casa de Misericórida de Juíz de Fora, Juiz de Fora, Minas Gerais
  - Associação Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Irmandade Santa Casa de Misericórdia de Marília, Marília, São Paulo